CLINICAL TRIAL: NCT06145867
Title: A Feasibility Study Assessing the Acceptability, Adherence, and Safety of Photobiomodulation (PBM) Therapy and Objective Assessment Measures in Myalgic Encephalomyelitis (ME)
Brief Title: A Feasibility Study: Assessing Photobiomodulation in Myalgic Encephalomyelitis
Acronym: LightMEup
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Quadram Institute Bioscience (Other)
Collaborators: University of East Anglia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QIB02/2023
Record Dates: First submitted 2023-10-04; First posted 2023-11-24 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Myalgic Encephalomyelitis; Chronic Fatigue Syndrome
Keywords: me/cfs
MeSH Terms: conditions — Fatigue Syndrome, Chronic | interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PBM therapy (Experimental): All participants will use the 670 nm lamp for 2 minutes each morning for 14 days.
  Interventions: Other: Photobiomodulation therapy

INTERVENTIONS:
Other: Photobiomodulation therapy — deep red light therapy (670nm)

SUMMARY:
There is no cure or approved treatments for ME. Several causes have been implicated in ME, including poor mitochondrial function. Mitochondria are the powerhouse of cells, producing energy. Therefore, loss of mitochondrial function and reduced energy production could be an explanation for the debilitating chronic fatigue that defines ME.

The primary site of red light absorption in cells is the mitochondria. Mitochondrial red light absorption can boost energy production. Light therapy is already FDA approved for the treatment of acne, muscle and joint pain, arthritis, blood circulation issues and hair loss. This is the first study to trial the use of red light therapy in ME and results will help us understand if the use of red light therapy is accepted by ME patients.

In past clinical trials the monitoring of symptom reduction/increase in ME patients was mainly done using symptom questionnaires. These questionnaires have not been specifically developed for ME symptoms and therefore the reliability of results is poor. This study will be assessing the use of a new symptom questionnaire developed specifically for ME and will also be trialling the use of other tools to measure symptom reduction/increase.

In addition, this study will also trial the use of Mantal, an online remote research management portal. This is to improve accessibility of ME patients to research participation.

Each ME participants involvement in the study should take approximately 7 weeks. Involvement is split into four phases: 1) baseline, 2) intervention, 3) follow-up and 4) feedback.

Baseline assessments:

* Week one: complete a 27-item questionnaire on functional capacity (FUNCAP27) and online cognitive function tests
* Week two: participants are posted an activity monitor which they are to wear for seven days. Participants will complete a sleep diary (consensus sleep diary version E) for seven days

Intervention:

- Participants are posted the red lamp to use in their own homes during weeks three and four. Participants use the red lamp for two minutes, daily, each morning for a total of 14 days.

Follow-up:

* Weeks five and six
* Repeating the baseline assessments

Feedback:

- Participants are asked to complete an online questionnaire during week seven.

DETAILED DESCRIPTION:
The prevailing theory regarding mechanism of action of PBM is that by activating cytochrome c oxidase (CCO) it boosts mitochondrial ATP production, which, in turn, enhances the metabolic activity of the cell. This occurs simultaneously with the regulation of the reduction/oxidation (redox) state of the intracellular microenvironment favouring expression of genes associated with tissue regeneration and repair. Immune modulation and dampening or attenuation of pro-inflammatory responses ensures a coordinated regenerative effort. An alternate mechanism of action, independent of the absorption of red and near infrared light by CCO, proposes that by reducing the viscosity of interfacial water layers in the predominantly hydrophilic intramitochondrial space PBM increases the speed of rotation and activity of the mitochondrial rotary motor (ATP synthase) that results in increased ATP production. Irrespective of the exact biochemical mechanism of action, crucially, these processes take place in the absence of inciting tissue injury, photothermal effects, or photoacoustic effects.

While the underlying causes of ME/CFS are not know a consistent finding from metabolism-based studies is mitochondrial dysfunction and compromised energy metabolism characterised by high levels of oxidative stress and limited ATP production. Loss of mitochondrial function and compromised ATP production is therefore a plausible explanation for the debilitating chronic fatigue that defines ME/CFS. Based upon prior human studies demonstrating restored ATP production and function investigators hypothesise that PBM and 670nm red light exposure will, by increasing mitochondrial function in ME/CFS patients, improve their physical capacity and cognitive function.

The device that will be used to evaluate red light therapy in ME/CFS patients is an LED lamp that emits a spectrum of light in the red spectrum of visible light, peaking at 670 nm. This lamp was purchased from Planet Lighting Ltd, London, UK; LBT-PAR38-40. This lamp has the following specifications: 1) 40W output, 2) 60o beam angle, 3) 220-240V 50Hz input, 4) E27 base, 5) has a UK Conformity Assessed (UKCA) marking, 6) has CE certification, 7) is Restriction of Hazardous Substances Directive (RoHS) compliant, 8) has a 3 years warranty. It is important to note that this is not a medical device and will be marketed by Planet Lighting as an aid to general health wellbeing lamp for the general population. The Planet Lighting website advertising this product is currently being developed. The director from Planet Lighting has confirmed this in a letter.

Participants will be identified through the UK charity Invest in ME Research. Potential participants are those who have subscribed to the charity. The charity will email subscribers the study flyer and the participant invitation letter. The study flyer and participant invitation letter will include a link to the study specific website on Mantal. The homepage of the study website will contain a summary of the study and a link to the full participant information sheet which ME patients can either download and print or read online.

At the end of the full participant information sheet participants will be instructed on how to provide their informed consent if they wish to participate. Participants will be asked to click on the "register now" button on the homepage of the study website. When participants click on the register now button they will be taken through a series of statements for their consent. If participants consent to all of the statements they will then be taken to a sign up page where participants are able to register for the study with their first and last name and email address. They will be asked to provide a password for their account.

After participants have provided informed consent and created an account on the study website participants will be asked to complete a screening questionnaire on the study website. Participants who fulfil the eligibility criteria will receive a notification to inform them that they are eligible and have been enrolled onto the study. The notification also prompts participants to log in to Mantal to complete baseline study procedures. Participants who do not fulfil the eligibility criteria will be notified on the screen that they are unable to participate in the study at this time and will receive a QIB withdrawal letter via email.

Once participants are enrolled onto the study, participants will be asked to complete the "About You" questionnaire, which will collect information on the participants demographics and ME diagnosis.

Then participants will move onto baseline measures. The first baseline measure participants are asked to complete is the FUNCAP27 questionnaire, which assesses functional capacity. Participants will complete the FUNCAP27 questionnaire online through Mantal. Once participants have completed this questionnaire, they will then complete the battery of six online cognitive function assessments from NeurOn (https://neuropsychology.online) in the following order: 1) reaction time, 2a) word encoding, 2b) word retrieval, 3) trails A, 4) trails B, 5) digit span backwards and 6) fragmented letters. Participants will complete cognitive assessments online through Mantal. Participants can choose to either complete the FUNCAP27 questionnaire and the cognitive function assessments on the same day or on separate days. Participants are asked to try to complete as many of the cognitive function assessments as they feel able to. Before and after each cognitive function assessment participants are asked to rate their level of cognitive fatigue (from 1 to 10, 1 being the worst and 10 being the best) and asked if they feel well enough to complete the next cognitive function assessment. If participants answer no, then the battery of cognitive function assessments will be terminated for that participant. Participants will receive daily text or email reminders to complete the FUNCAP27 and NeurOn assessments. After participants have completed or terminated the cognitive function assessments they will be asked to provide their address for the research team to mail the GENEActiv wrist worn accelerometer monitor and instructions to participants. Participants will be asked to complete an equipment disclaimer form online prior to wearing the accelerometer. Participants will be asked to wear these monitors immediately upon receipt for a total of seven days. Participants will receive daily automatic text reminders sent out by Mantal to wear the monitor. Participants are asked to enter the date they start wearing the monitor onto the study portal. Once participants have confirmed they are wearing the monitor, participants will be able to complete the morning and evening entries of the consensus sleep diary version E (CSD-E) for the seven days they are wearing the monitor. Participants will receive daily text reminders (automatically sent out by Mantal) to complete the CSD-E morning and evening entries. Seven days from the date they start wearing the monitor participants will receive a text reminder (automatically sent out by Mantal) to take off the monitors and to post them back to the research team using the prepaid envelope. Participants who are housebound are asked to contact the research team to arrange a courier to collect the GENEActiv accelerometer from participants homes. Participants will receive a text reminder daily until the research team has received the monitor. The PI will download the raw data from the devices internal memory and perform a quality control (QC) check that the monitor has worked and recorded activity for 7 days. If the monitor has not worked participants will be requested to repeat the wear of the monitor and completing the CSD-E.

Once the activity monitor data has passed the QC the red lamp (Planet Lighting Ltd, London, UK) will be posted to participants with instructions for use. Participants will complete an online donated equipment disclaimer form before using the lamps. Participants will be asked to use this lamp for 2 minutes, daily (between 9:00 and 11:00), for a total of 2 weeks. Participants will receive daily text reminders at 8:30 to use the lamp. Participants will be asked to log on to mantal each day and record whether they have managed to use the lamp that day. After using the lamp for 2 weeks participants will be asked to return the lamp back to the research team using the prepaid postage labels. Participants who are housebound are asked to contact the research team to arrange a home collection via courier.

Once participants have finished the intervention, they are asked to complete the FUNCAP27 questionnaire, NeurOn assessments, wear the GENEActiv monitor and the complete the CSD-E. This will be undertaken following the same protocol as the baseline measures. Once the research team has received the monitors in the post participants will be asked to complete a feedback questionnaire via Mantal.

The end of the study will be when the last participant has completed the feedback questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have received an ME diagnosis from primary or secondary care
* must be able to understand the requirements of the study and provide informed consent.
* must live in the UK

Exclusion Criteria:

* Participants who have received one or more of the following diagnoses: 1) any illness other than ME/CFS that has fatigue as a symptom (e.g. multiple sclerosis or inherited mitochondrial disease), 2) any illness with cognitive defects (e.g. alzheimer's disease, dementia), 3) any proliferative disease (e.g. cancer), 4) any surface bacterial/fungal infection (e.g. blepharitis)
* Participants who have altered their medication within the last 4 weeks
* Participants who have made major dietary alterations within the last 4 weeks
* Participants who have underwent surgery requiring general anaesthetic within the last 6 months
* Participants who have broken/fractured/torn any bones or ligaments within the last 6 months
* Participants who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Compliance of PBM therapy in ME patients. | Week 3 and 4
  Compliance will be measured when participants log in daily into Mantal study portal to confirm the use of the lamp during the 14 days from week 3 to 4.
Acceptance of PBM therapy in ME patients. | Week 7
  Acceptance will be measured at week 7 using the Feedback questionnaire which will ask about ease of setting up the red lamp (PBM), ease of use during the 14 day intervention and future use of lamp. The responses are binary (YES or NO). Greater number of YES responses compared to NO responses will indicate that PBM therapy was acceptable in ME patients.
Safety of PBM therapy in ME patients. | Week 3, 4, and 7
  Self-reported adverse reaction or event by participants to the red (PBM) lamp will be used to measure safety. Safety will be measured at week 3 (start of intervention) through week 4 (at the end of intervention) and at week 7 (feedback questionnaire). The severity of the adverse event will be reported using the University of East Anglia and Norfolk and Norwich University Hospitals SOP 205 guidelines. Safety will be reported as mild, moderate, or severe. PBM therapy in ME patients will be regarded safe when severity of self-reported adverse reaction is no greater than mild in severity.

SECONDARY OUTCOMES:
Compliance of the GENEActiv accelerometers in ME patients | Week 2
  Compliance will be measured with daily completion of the consensus sleep diary version E during the 7-day intervention at week 2.
Acceptance of the GENEActiv accelerometers in ME patients | Week 2 and week 7
  Acceptance will be measured at week 2 when participants initially sign into Mantal study portal at the start of intervention and at week 7 with the Feedback questionnaire which will ask about ease of wearing the accelerometer. The responses are binary (YES or NO). Greater number of YES responses compared to NO responses will indicate that the GENEActiv accelerometers was acceptable in ME patients.
Safety of GENEActiv accelerometers in ME patients. | Week 2, 6, and 7
  Self-reported adverse reaction or event by participants to the accelerometer. Safety will be measured at week 2 (during intervention), at week 6 (follow-up phase) and at week 7 (feedback questionnaire). The severity of the adverse event will be reported using the University of East Anglia and Norfolk and Norwich University Hospitals SOP 205 guidelines. Safety will be reported as mild, moderate, or severe. GENEActiv accelerometers in ME patients will be regarded safe when severity of self-reported adverse reaction is no greater than mild in severity.
Changes in NeurOn (online cognitive function assessments) completion rates in ME patients. | Week 1 and 5
  Comparison of the completion rates in NeurOn will be assessed at baseline (week 1) and follow up visit (week 5).
Acceptability of NeurOn in ME patients. | Week 7
  Feedback questionnaire at week 7 regarding NeurON (online cognitive function assessments) will be used to measure the ease of using an online cognitive function test and the acceptability of the number of assessments that were administered during the study.
Acceptability of FUNCAP27 in ME patients. | Week 7
  Feedback questionnaire at week 7 regarding FUNCAP27 (quantitative assessment of functional capacity) will be use to measure the acceptability of the length of FUNCAP27 assessment and ability to understand the questions in FUNCAP27.
Compliance of the consensus sleep diary version E (CSD-E) in ME patients. | Week 2
  Number of completed daily sleeping diaries submitted during the 7 day intervention (week 2)
Acceptability of the consensus sleep diary version E (CSD-E) in ME patients. | Week 7.
  Feedback questionnaire at week 7 regarding consensus sleep diary version E will be used to measure the acceptability by assessing the ease of use and frequency of sleep diary documentation (day and evenings).
Acceptability of Mantal in ME patients. | week 7
  Feedback questionnaire at week 7 regarding Mantal (online study and participant management tool) will be used to measure acceptability by assess the ease of using Mantal study portal and use of online informed consent procedure, and the notifications sent by Mantal.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Carding, PhD, Principal Investigator — Quadram Institute Bioscience
Locations (1):
- Quadram Institute Bioscience, Norwich, Norfolk, United Kingdom

IPD SHARING:
Plan to Share IPD: No